CLINICAL TRIAL: NCT05326789
Title: Coronary and Cerebral Perfusion Optimization in Cardiac Arrest: A Feasibility and Physiological Study
Acronym: CC-POCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2677
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Arrest
Keywords: REBOA; ROSC; Cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: single-center, single-arm, open (unblinded), feasibility, experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- interventional (Experimental): 20 patients with inclusion criteria and without exclusion criteria will be entered in the interventional arm attempting to use REBOA during non-traumatic cardiac arrest.
  Interventions: Device: REBOA catheter

INTERVENTIONS:
Device: REBOA catheter — balloon occlusion of the aorta during cardiac arrest to optimize coronary and cerebral perfusion.
  Other Names: resuscitative endovascular balloon occlusion of the aorta

SUMMARY:
Our general objective, during this study, is to evaluate the feasibility and potential physiological benefits of using REBOA (resuscitative endovascular balloon occlusion of the aorta) CPR (cardiopulmonary resuscitation) for patients presenting with a cardiac arrest to a community hospital. This would represent the first step for doing a larger, randomized clinical trial on the use of REBOA in non-traumatic cardiac arrest.

DETAILED DESCRIPTION:
Primary objective: Validate the feasibility of using REBOA in a community hospital setting during cardiac arrest as an adjunct to ACLS (advances cardiac life support) . This will be done by measuring time to REBOA placement and successful inflation. Furthermore, we will also document any REBOA related complications.

Secondary objectives: Evaluate the potential physiological benefits of REBOA for human subjects in NTCA (non traumatic cardiac arrest) that are not responding to standard ACLS.

Study Design and Methodology Trial design The trial is a single-center, single-arm, open (unblinded), feasibility, experimental study.

Study Duration The study is expected to begin in winter 2022 and last approximately 12 months. Population studied The population studied will be patients in non-traumatic cardiac arrest at Santa Cabrini Hospital, aged 18-75 years old.

Patients presenting with a witnessed cardiac arrest (out of hospital cardiac arrest (OHCA) or in hospital cardiac arrest (IHCA)) and in which ACLS was performed for at least 15 minutes or BLS for at least 30 minutes and for no more than 60 minutes will be evaluated for eligibility to participate in the study.

Number of patients 20

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged 18-75 years old
* Suspected reversible cause of cardiac arrest (except for trauma), with one of any of the following prognostic signs30

  * Reactive pupils
  * Agonal breathing
  * EtCO2>10 mmHg
  * Any cardiac activity on bedside echocardiogram
* Body habitus accommodating automated Lund University Cardiac Arrest System (LUCAS)
* Level of care includes CPR, or unable to obtain level of care (if possible, validate with relative)
* More than 15 minutes of ACLS with no ROSC or more than 30 minutes of BLS with no ROSC

Exclusion Criteria:

* Transfer accepted for ECPR

  * History of severe dementia
  * Advance Medical Directives against resuscitation
  * History of aortic pathology or surgery
  * LUCAS not compatible with the patient's body habitus
  * Pregnancy
  * Any illness resulting in loss of independent living capacity
  * Severe cardiopulmonary disease
  * Aortic dissection, aortic aneurysm, tension pneumothorax or tamponade seen on TEE/TTE
  * Strangulation
  * Suspected intracerebral hemorrhage
  * Accidental hypothermia
  * More than 60 minutes of resuscitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
success rate and time of REBOA inflation during non-traumatic arrest in a community hospital | 1 year
  ● Feasibility of intra-arrest REBOA catheter placement and zone 1 inflation in NTCA in a community hospital setting

SECONDARY OUTCOMES:
blood pressure | 0-15 min per study over a year
  * Systolic blood pressure (Pre balloon occlusion, Post balloon occlusion 30sec, 1min, 5min, 10min, 15min)
  * Diastolic blood pressure (Pre balloon occlusion, Post balloon occlusion 30sec, 1min, 5min, 10min, 15min)
ETCO2 | 0-15 min per study over a year
  (Pre balloon occlusion, Post balloon occlusion 30sec, 1min, 5min, 10min, 15min)
cerebral saturation | 0-15 min per study over a year
  (Pre balloon occlusion, Post balloon occlusion 30sec, 1min, 5min, 10min, 15min)
ROSC | 0-30 min per study over a year
  return of spontaneous circulation
TEE-guided REBOA positioning | 5 minutes per study over 1 year
  success rate of determining REBOA placement by trans esophageal echocardiography
7 day survival | 7 days over a year
  follow up to 7 days

IPD SHARING:
Plan to Share IPD: Undecided